CLINICAL TRIAL: NCT06588946
Title: The Effect of Exogenous Β-OHB Supplementation on Cerebral Blood Flow and Functional Brain Characteristics in Adults with Subjective Cognitive Decline
Brief Title: Β-OHB Supplementation and Brain Health in Older Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Jeremy Walsh, Assistant Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 05992572
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Subjective Cognitive Decline
Keywords: early-stage dementia; ketone monoester supplementation; cerebral blood flow; cognition; resting state functional magnetic resonance imaging; placebo
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone monoester (KME) supplement (Experimental): Participants will be instructed to consume a ketone monoester (KME) supplement prior to each meal (3x/day) for 14 days.
  Interventions: Dietary Supplement: Ketone monoester (KME) supplement
- Placebo supplement (Placebo Comparator): Participants will be instructed to consume a bottle of placebo supplement prior to each meal (3x/day) for 14 days.
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Ketone monoester (KME) supplement — 15g of a KME supplement orally consumed 3x daily for 14 days. This dosing protocol raises plasma β-OHB consistently during the waking hours. Oral KME will be provided in opaque bottles labelled A or B to maintain condition blinding. Each bottle will contain a drink providing 15g of a KME supplement: [R]-3-hydroxybutyl [R]-3-hydroxybutyrate (ΔG®, TDeltaS, Oxford, UK).
  Other Names: [R]-3-hydroxybutyl [R]-3-hydroxybutyrate (ΔG®, TDeltaS, Oxford, UK)
  Arms: Ketone monoester (KME) supplement
Dietary Supplement: Placebo supplement — 50mL taste-match inert calorie-free placebo drink orally consumed 3x daily for 14 days. Oral placebo will be provided in opaque bottles labelled A or B to maintain condition blinding.
  Arms: Placebo supplement

SUMMARY:
The goal of this randomized placebo controlled crossover trial is investigate the effects of short-term ketone monoester (KME) supplementation to brain function in older adults with subjective cognitive decline. We will test the hypothesis that KME supplementation will increase cerebral blood flow and improve resting-state functional connectivity in the brain compared to placebo supplementation in older adults with subjective cognitive decline.

Participants will be randomly assigned to either placebo of KME supplementation for 14 days. Following a washout period, participants will complete the alternate condition for 14 days. Outcome measures will be assessed before and after each intervention period.

DETAILED DESCRIPTION:
In this randomized placebo-controlled crossover double-blind designed clinical trial, 48 adults with SCD (50% female; aged 55 to 75 years old) will be allocated to a ketone monoester (KME) or placebo condition in random order (e.g., A-B or B-A), stratified by sex. Participants will be recruited from the local community through McMaster University, the local Alzheimer Society, and community outreach.

In total, participants will be asked to complete 5 visits. Data will be collected at a single site in Hamilton, Ontario associated with McMaster University. All interested individuals will complete an eligibility screening study visit (Visit 1) to establish inclusion/exclusion. Written, informed consent will be obtained before data collection. Demographic information and medical history will be collected at the beginning of Visit 1 to obtain information regarding medication use, medical history, age, years of education, and sex and gender-based variables. This information will be collected using a participant history questionnaire and the GENESIS-PRAXY questionnaire. Participants will also be introduced to the lab and the different tests that we will run during the experimental visits. Data will be collected at two time points for each condition: 1) Pre-intervention (Visits 2 & 4: baseline); and post-intervention (Visits 3 & 5: following 14-day intervention). In a randomized crossover design, participants will be randomly allocated to a condition (placebo or KME) for a 14-day intervention. Participants will then undergo a washout period, afterwhich participants will be complete the alternate condition including baseline data collection (Visit 4) and post-intervention visit (Visit 5) after the second 14-day intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Being objectively cognitively normal as determined by a Montreal Cognitive Assessment (MoCA) score ≥26 with independent living and ambulating
* SCD will be determined using the Prospective-Retrospective Memory Questionnaire (PRMQ) following the SCD Initiative Working Group framework

Exclusion Criteria:

* A diagnosis of mild cognitive impairment, dementia, or psychiatric and/or mood disorders (e.g., major depression)
* MoCA score <26
* Diagnosis of cardiometabolic disease (e.g., hypertension, type 2 diabetes)
* Obesity (BMI >30 kg/m2)
* History of heart attack or stroke
* History of smoking
* Currently following a ketogenic diet or taking ketogenic supplements
* Having MRI contraindications
* Participants with literacy, visual, hearing, and/or speech issues, as well as individuals who are not proficient in English will not be eligible for this trial

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Global cerebral blood flow (gCBF) | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  Measured by magnetic resonance imaging (MRI) under resting, normocapnic conditions. Arterial flow measurement will be performed using a phase contrast flow sensitizing MRI pulse sequence. Cross-sectional areas and mean blood flow of the carotid and vertebral arteries will be measured, with total blood flow in all four vessels equaling global CBF.
Resting-state functional connectivity | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  A resting state functional magnetic resonance imaging (rsfMRI) scan will be performed eyes closed using a gradient echo EPI sequence. The temporal and regional co-activation of brain regions in the resting state provide a measure of functional connectivity in the brain. rsfMRI data will be analyzed to measure global whole-brain functional connectivity and within localized brain regions of interest.

SECONDARY OUTCOMES:
Cognitive testing | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  A battery of computerized validated psychometric tests will be used, including: the Mnemonic similarities task (MST) to assess hippocampal-dependent learning and memory, the Stroop colour-word task to assess processing speed, working memory, attention, and inhibitory control, and a shortened version of the Odd-One-Out test to measure working memory and executive function. A non-computerized dual-task test will be performed to assess the multitasking ability of walking while performing another cognitive task.
Microstructural white matter health | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  Dual spin echo, echo-planar imaging (EPI) diffusion tensor imaging (DTI) sequence collected by magnetic resonance imaging (MRI) to assess brain white matter microstructural integrity.
Cerebrovascular reactivity | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  The phase contrast flow sensitizing MRI pulse and resting state functional MRI sequences will both be repeated while participants undergo an elevated CO2 breathing task. Cerebrovascular function will be calculated from the stimulus-response relationship between PaCO2 and (1) phase contrast: cross sectional areas of the internal carotid and vertebral arteries, and (2) rsfMRI: % change BOLD/mmHg.
Blood-borne biomarkers | Baseline and post-intervention (i.e., 14-days later) for both KME and placebo conditions
  A venous blood sample will be collected to assess circulating concentrations of various hormones and metabolites (e.g., brain-derived neurotrophic factor [BDNF]) that relate to brain health, metabolism, and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Walsh, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers from a reputable institution who wish to access the data may submit a request to the Principal Investigator.

REFERENCES:
- [Background] 2023 Alzheimer's disease facts and figures. Alzheimers Dement. 2023 Apr;19(4):1598-1695. doi: 10.1002/alz.13016. Epub 2023 Mar 14. PMID 36918389
- [Background] Al-Khazraji BK, Buch S, Kadem M, Matushewski BJ, Norozi K, Menon RS, Shoemaker JK. Protocol-dependence of middle cerebral artery dilation to modest hypercapnia. Appl Physiol Nutr Metab. 2021 Sep;46(9):1038-1046. doi: 10.1139/apnm-2021-0220. Epub 2021 Jun 17. PMID 34139129
- [Background] Alzheimer's Society of Canada. Rising Tide: The Impact of Dementia on Canadian Society. 2010; ISBN 978-0-9733522-2-1
- [Background] Cunnane SC, Courchesne-Loyer A, Vandenberghe C, St-Pierre V, Fortier M, Hennebelle M, Croteau E, Bocti C, Fulop T, Castellano CA. Can Ketones Help Rescue Brain Fuel Supply in Later Life? Implications for Cognitive Health during Aging and the Treatment of Alzheimer's Disease. Front Mol Neurosci. 2016 Jul 8;9:53. doi: 10.3389/fnmol.2016.00053. eCollection 2016. PMID 27458340
- [Background] Cunnane SC, Trushina E, Morland C, Prigione A, Casadesus G, Andrews ZB, Beal MF, Bergersen LH, Brinton RD, de la Monte S, Eckert A, Harvey J, Jeggo R, Jhamandas JH, Kann O, la Cour CM, Martin WF, Mithieux G, Moreira PI, Murphy MP, Nave KA, Nuriel T, Oliet SHR, Saudou F, Mattson MP, Swerdlow RH, Millan MJ. Brain energy rescue: an emerging therapeutic concept for neurodegenerative disorders of ageing. Nat Rev Drug Discov. 2020 Sep;19(9):609-633. doi: 10.1038/s41573-020-0072-x. Epub 2020 Jul 24. PMID 32709961
- [Background] Frei M, Berres M, Kivisaari SL, Henzen NA, Monsch AU, Reinhardt J, Blatow M, Kressig RW, Krumm S. Can you find it? Novel oddity detection task for the early detection of Alzheimer's disease. Neuropsychology. 2023 Oct;37(7):717-740. doi: 10.1037/neu0000859. Epub 2022 Oct 6. PMID 36201797
- [Background] GBD 2019 Dementia Forecasting Collaborators. Estimation of the global prevalence of dementia in 2019 and forecasted prevalence in 2050: an analysis for the Global Burden of Disease Study 2019. Lancet Public Health. 2022 Feb;7(2):e105-e125. doi: 10.1016/S2468-2667(21)00249-8. Epub 2022 Jan 6. PMID 34998485
- [Background] Han YM, Bedarida T, Ding Y, Somba BK, Lu Q, Wang Q, Song P, Zou MH. beta-Hydroxybutyrate Prevents Vascular Senescence through hnRNP A1-Mediated Upregulation of Oct4. Mol Cell. 2018 Sep 20;71(6):1064-1078.e5. doi: 10.1016/j.molcel.2018.07.036. Epub 2018 Sep 6. PMID 30197300
- [Background] Harris JA, Benedict FG. A Biometric Study of Human Basal Metabolism. Proc Natl Acad Sci U S A. 1918 Dec;4(12):370-3. doi: 10.1073/pnas.4.12.370. No abstract available. PMID 16576330
- [Background] Iadecola C. The pathobiology of vascular dementia. Neuron. 2013 Nov 20;80(4):844-66. doi: 10.1016/j.neuron.2013.10.008. PMID 24267647
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Shaw LM, Aisen PS, Weiner MW, Petersen RC, Trojanowski JQ. Hypothetical model of dynamic biomarkers of the Alzheimer's pathological cascade. Lancet Neurol. 2010 Jan;9(1):119-28. doi: 10.1016/S1474-4422(09)70299-6. PMID 20083042
- [Background] Jensen NJ, Nilsson M, Ingerslev JS, Olsen DA, Fenger M, Svart M, Moller N, Zander M, Miskowiak KW, Rungby J. Effects of beta-hydroxybutyrate on cognition in patients with type 2 diabetes. Eur J Endocrinol. 2020 Feb;182(2):233-242. doi: 10.1530/EJE-19-0710. PMID 31821157
- [Background] Jessen F, Wiese B, Bachmann C, Eifflaender-Gorfer S, Haller F, Kolsch H, Luck T, Mosch E, van den Bussche H, Wagner M, Wollny A, Zimmermann T, Pentzek M, Riedel-Heller SG, Romberg HP, Weyerer S, Kaduszkiewicz H, Maier W, Bickel H; German Study on Aging, Cognition and Dementia in Primary Care Patients Study Group. Prediction of dementia by subjective memory impairment: effects of severity and temporal association with cognitive impairment. Arch Gen Psychiatry. 2010 Apr;67(4):414-22. doi: 10.1001/archgenpsychiatry.2010.30. PMID 20368517
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886
- [Background] Jessen F, Amariglio RE, Buckley RF, van der Flier WM, Han Y, Molinuevo JL, Rabin L, Rentz DM, Rodriguez-Gomez O, Saykin AJ, Sikkes SAM, Smart CM, Wolfsgruber S, Wagner M. The characterisation of subjective cognitive decline. Lancet Neurol. 2020 Mar;19(3):271-278. doi: 10.1016/S1474-4422(19)30368-0. Epub 2020 Jan 17. PMID 31958406
- [Background] Krikorian R, Shidler MD, Dangelo K, Couch SC, Benoit SC, Clegg DJ. Dietary ketosis enhances memory in mild cognitive impairment. Neurobiol Aging. 2012 Feb;33(2):425.e19-27. doi: 10.1016/j.neurobiolaging.2010.10.006. Epub 2010 Dec 3. PMID 21130529
- [Background] Li M, Zheng G, Zheng Y, Xiong Z, Xia R, Zhou W, Wang Q, Liang S, Tao J, Chen L. Alterations in resting-state functional connectivity of the default mode network in amnestic mild cognitive impairment: an fMRI study. BMC Med Imaging. 2017 Aug 16;17(1):48. doi: 10.1186/s12880-017-0221-9. PMID 28814282
- [Background] McCrimmon RJ, Ryan CM, Frier BM. Diabetes and cognitive dysfunction. Lancet. 2012 Jun 16;379(9833):2291-9. doi: 10.1016/S0140-6736(12)60360-2. Epub 2012 Jun 9. PMID 22683129
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Mujica-Parodi LR, Amgalan A, Sultan SF, Antal B, Sun X, Skiena S, Lithen A, Adra N, Ratai EM, Weistuch C, Govindarajan ST, Strey HH, Dill KA, Stufflebeam SM, Veech RL, Clarke K. Diet modulates brain network stability, a biomarker for brain aging, in young adults. Proc Natl Acad Sci U S A. 2020 Mar 17;117(11):6170-6177. doi: 10.1073/pnas.1913042117. Epub 2020 Mar 3. PMID 32127481
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Nation DA, Sweeney MD, Montagne A, Sagare AP, D'Orazio LM, Pachicano M, Sepehrband F, Nelson AR, Buennagel DP, Harrington MG, Benzinger TLS, Fagan AM, Ringman JM, Schneider LS, Morris JC, Chui HC, Law M, Toga AW, Zlokovic BV. Blood-brain barrier breakdown is an early biomarker of human cognitive dysfunction. Nat Med. 2019 Feb;25(2):270-276. doi: 10.1038/s41591-018-0297-y. Epub 2019 Jan 14. PMID 30643288
- [Background] Neudorf H, Islam H, Falkenhain K, Oliveira B, Jackson GS, Moreno-Cabanas A, Madden K, Singer J, Walsh JJ, Little JP. Effect of the ketone beta-hydroxybutyrate on markers of inflammation and immune function in adults with type 2 diabetes. Clin Exp Immunol. 2024 Mar 12;216(1):89-103. doi: 10.1093/cei/uxad138. PMID 38195093
- [Background] Petrella JR, Sheldon FC, Prince SE, Calhoun VD, Doraiswamy PM. Default mode network connectivity in stable vs progressive mild cognitive impairment. Neurology. 2011 Feb 8;76(6):511-7. doi: 10.1212/WNL.0b013e31820af94e. Epub 2011 Jan 12. PMID 21228297
- [Background] Roy M, Edde M, Fortier M, Croteau E, Castellano CA, St-Pierre V, Vandenberghe C, Rheault F, Dadar M, Duchesne S, Bocti C, Fulop T, Cunnane SC, Descoteaux M. A ketogenic intervention improves dorsal attention network functional and structural connectivity in mild cognitive impairment. Neurobiol Aging. 2022 Jul;115:77-87. doi: 10.1016/j.neurobiolaging.2022.04.005. Epub 2022 Apr 12. PMID 35504234
- [Background] Shimazu T, Hirschey MD, Newman J, He W, Shirakawa K, Le Moan N, Grueter CA, Lim H, Saunders LR, Stevens RD, Newgard CB, Farese RV Jr, de Cabo R, Ulrich S, Akassoglou K, Verdin E. Suppression of oxidative stress by beta-hydroxybutyrate, an endogenous histone deacetylase inhibitor. Science. 2013 Jan 11;339(6116):211-4. doi: 10.1126/science.1227166. Epub 2012 Dec 6. PMID 23223453
- [Background] Smith G, Della Sala S, Logie RH, Maylor EA. Prospective and retrospective memory in normal ageing and dementia: a questionnaire study. Memory. 2000 Sep;8(5):311-21. doi: 10.1080/09658210050117735. PMID 11045239
- [Background] Stark SM, Kirwan CB, Stark CEL. Mnemonic Similarity Task: A Tool for Assessing Hippocampal Integrity. Trends Cogn Sci. 2019 Nov;23(11):938-951. doi: 10.1016/j.tics.2019.08.003. Epub 2019 Oct 6. PMID 31597601
- [Background] Stroop, JR. Studies of interference in serial verbal reactions. J Exp Psychol. 1935;18:643-662. doi: 10.1037/h0054651
- [Background] Svart M, Gormsen LC, Hansen J, Zeidler D, Gejl M, Vang K, Aanerud J, Moeller N. Regional cerebral effects of ketone body infusion with 3-hydroxybutyrate in humans: Reduced glucose uptake, unchanged oxygen consumption and increased blood flow by positron emission tomography. A randomized, controlled trial. PLoS One. 2018 Feb 28;13(2):e0190556. doi: 10.1371/journal.pone.0190556. eCollection 2018. PMID 29489818
- [Background] Walsh JJ, Caldwell HG, Neudorf H, Ainslie PN, Little JP. Short-term ketone monoester supplementation improves cerebral blood flow and cognition in obesity: A randomized cross-over trial. J Physiol. 2021 Nov;599(21):4763-4778. doi: 10.1113/JP281988. Epub 2021 Oct 4. PMID 34605026
- [Background] Walsh JJ, Neudorf H, Little JP. 14-Day Ketone Supplementation Lowers Glucose and Improves Vascular Function in Obesity: A Randomized Crossover Trial. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1738-e1754. doi: 10.1210/clinem/dgaa925. PMID 33367782